CLINICAL TRIAL: NCT06846021
Title: Single-cell Immunomics Research on the Onset and Different Outcomes in Patients with Ankylosing Spondylitis
Brief Title: Integral Single-cell Landscape of Immunological Hallmarks for Ankylosing Spondylitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fujian Provincial Hospital (Other)
Responsible Party: Principal Investigator, Dianshan Ke, Principal Investigator, Fujian Provincial Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: K2022-09-055
Record Dates: First submitted 2025-02-12; First posted 2025-02-25 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-02

CONDITIONS: Ankylosing Spondylitis
MeSH Terms: conditions — Spondylitis, Ankylosing

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- The investigators performed single-cell RNA sequencing based on PBMCs (Experimental)
  Interventions: Other: Disease status

INTERVENTIONS:
Other: Disease status — According to the disease status, patients are divided into four groups including healthy donors, initial patients with high activity, patients with deformities and patients with clinical remission

SUMMARY:
Three HLA-B27-positive health donors (HDs) with matching age were enrolled via genetic screening, and fourteen AS patients were recruited at Fujian provincial hospital from May to July 2021. All AS patients satisfied the modified New York (NY) criteria, and the categorization of three disease groups (EA, LD and RM) was according to clinical hallmarks and imaging evidences. The five patients in the EA group were in the early stage of disease, showing obvious symptoms, and had not yet received standard treatments, including various NSAIDs and DMARDs. The five patients in the LD group were all disabled, and confirmed by radiographic evidence of structural damage in hip joints and spinal deformity. The four patients in the RM group received standardized treatment under the guidance of specialist doctors, and maintained clinical remission and normal laboratory indicators for over six months. Patients in both EA and RM groups were confirmed to have no structural damage or deformities by radiographic evidences.

ELIGIBILITY:
Inclusion Criteria:

Clinical diagnosis of ankylosing spondylitis Clinical hallmarks and imaging evidences

Exclusion Criteria:

Pregnant patients Other diseases, tumors and injuries

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2021-05-17 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-08-25 (Actual)

PRIMARY OUTCOMES:
Assessment of the immunological characteristics regarding the onset and outcomes of ankylosing-spondylitis patients relying on single-cell transcriptomics analysis for four groups of subjects (including health donors and patients in early active stage, l | 8 months

CONTACTS AND LOCATIONS:
Locations (1):
- Orthopedic Outpatient Room, Fuzhou, China